CLINICAL TRIAL: NCT01266538
Title: Epidemiologic, Clinical, Endoscopic and Histological Database of Patients With Inflammatory Bowel Disease (IBD)
Brief Title: Inflammatory Bowel Disease(IBD)Database
Acronym: IBD
Status: Not yet recruiting | Type: Observational
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Dr. Iris Dotan, Tel-Aviv Sourasky Medical Center
Other Study IDs: TASMC-10-ID-467-CTIL
Record Dates: First submitted 2010-12-23; First posted 2010-12-24 (Estimated); Last update posted 2010-12-24 (Estimated); Status verified 2010-12

CONDITIONS: Inflammatory Bowel Disease
MeSH Terms: conditions — Inflammatory Bowel Diseases

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood serum, gastrointestinal biopsies, fecal samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- IBD patients: Patients diagnosed with Inflammatory Bowel Disease (IBD)
- patients after a Large Bowel Resection: Patients after a Large Bowel Resection, with or without a pouch.
- Control group: Family members of IBD patients, Patients with Irritable Bowel Syndrome (IBS), Fap (familial polyposis)patients after a large bowel resection, Patient performing screening endoscopy

SUMMARY:
This will be a comprehensive epidemiological, clinical, endoscopic and histological database for inflammatory bowel diseases patients in our medical center that will further provide clinical and basic investigations.

DETAILED DESCRIPTION:
Inflammatory bowel diseases (IBD), which include Crohn's disease (CD), ulcerative colitis (UC), undefined IBD and pouchitis (in patients who required IPAA for their colitis) affects about two million people in the world. At this time there is no definitive cure and current treatment is aimed at managing the symptoms and inflammation that accompany these diseases. These diseases are predominantly chronic, and patients may experience various gastrointestinal symptoms depending on the location, nature, and extent of their disease. Both genetic and environmental factors play etiological roles. The overall goal of our research is to understand the etiology and course of these diseases in order to prevent and to manage cases more effectively. In order to do so we are aiming at building a comprehensive database that will include detailed clinical data conjoined with dedicated research information and collection of biological specimens that will target the gut epithelium immune system, the microbiota and specific genetic risk factors.

ELIGIBILITY:
Inclusion Criteria:

Diagnosis of IBD Regular treatment and follow up in Tel Aviv Sourasky medical center Fap (familial polyposis)patients after a large bowel resection, as controls Family members of IBD patients as controls Patients with Irritable Bowel Syndrome (IBS), as controls -

Exclusion Criteria:

pregnancy age<18 years

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 1. Cases: Patients diagnosed with Inflammatory Bowel Disease (IBD) attending the departement of Gastroenterology (Tel Aviv Sourasky Medical Center) for a regular follow up / treatment.
  2. Controls:Family members of IBD patients, Patients with Irritable Bowel Syndrome (IBS), Fap (familial polyposis)patients after a large bowel resection, Patient performing screening endoscopy
     --------------------------------------------------------------------------------
Sampling Method: Probability Sample
Enrollment: 2500 (Estimated)
Dates: Start 2011-01; Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
flactuations in gastrointestinal inflammation | ongoing, up to 4 times a year

SECONDARY OUTCOMES:
development of IBD-related morbidity and complications over time | ongoing, up to 4 times a year

CONTACTS AND LOCATIONS:
Overall Officials: Iris Dotan, MD PhD, Principal Investigator — Tel-Aviv Sourasky Medical Center
Locations (1):
- Tel Aviv Sourasky Medical Center, Tel Aviv, Israel